CLINICAL TRIAL: NCT06825429
Title: Group Exercise in Cancer Patients Under Active Treatment: Feasibility Pilot Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EFG 21/22
Record Dates: First submitted 2025-01-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-12

CONDITIONS: Neoplastic Disease
MeSH Terms: conditions — Neoplasms | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Single-centre, uncontrolled interventional feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECOG 0-1 (Experimental): Each 45-minute session includes an initial relaxation/stretching phase, simple aerobic exercises, muscle strengthening exercises, balance exercises and will be led by a physiotherapist
  Interventions: Procedure: exercise programme for group with ECOG 0-1
- ECOG 2 (Experimental): The exercises proposed to the group with ECOG 2 will be less intense and less difficult with the aim of adapting the activity to patients with a lower performance status
  Interventions: Procedure: exercise programme for ECOG 2 group

INTERVENTIONS:
Procedure: exercise programme for group with ECOG 0-1 — exercise programme for group with ECOG 2
  Arms: ECOG 0-1
Procedure: exercise programme for ECOG 2 group — this intervention shall be proportionated to the ECOG status of the group
  Arms: ECOG 2

SUMMARY:
The aim of this study to investigate the feasibility in hospital reality, of a group exercise program for oncology patients under active treatment and evaluate its impact on some outcomes considered relevant from both clinical and subjective point of view.

DETAILED DESCRIPTION:
The intervention will consist of EFG sessions lasting 45 minutes each, twice a week for 12 weeks to be carried out in the gym of the Rehabilitation Day Hospital.

Each 45-minute session includes an initial relaxation/stretching phase, simple aerobic exercises, muscle strengthening exercises, balance exercises, and will be led by a physiotherapist. The exercises proposed to the group with ECOG 2 will be less intense and of less difficulty with the aim of adapting the activity to patients with a lower performance status (see appendix 4.5, V2, 07/10/2024). The groups will consist of a minimum of five patients and a maximum of ten. Patients will also be stimulated to perform physical activity at home to a total of 150 minutes per week. Patients will be assessed at baseline (T0), at the end of the intervention (T1,12 weeks) and 6 months after the start of the intervention (T2).

ELIGIBILITY:
Inclusion Criteria:

* neoplastic tumor
* age>= 18
* prognosis> 12 months
* ECOG <=2
* Walking with/ without aids
* clinically stable
* signed informed consent
* Patients with bone metastases with ECOG from 0-1 suitable results

Exclusion Criteria:

* sensory deficits who cannot perform physical exercise
* cognitive impairment that compromises collaboration and questionnaire filling
* patients with pathologies (e.g. neurological, psychiatric) that do not allow the obtaining of valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
adherence to the group exercise programme | through study completion, an average of 2 years
  overall adherence to the group exercise programme > 40%
Frequency | through study completion, an average of 2 years
  The frequency of at least 70% of the exercise sessions foreseen by the programme.

SECONDARY OUTCOMES:
QoL | through study completion, an average of 2 years
  Questionnaire in which patients have to describe quality of life during study treatment
tolerance to effort | through study completion, an average of 2 years
  The effect of the EFG program on mood tone and physical function

CONTACTS AND LOCATIONS:
Overall Officials: Besa Kopliku, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna